CLINICAL TRIAL: NCT00923130
Title: A Phase II Multi-Center Study of Bevacizumab in Combination With Ixabepilone in Subjects With Advanced Renal Cell Carcinoma
Brief Title: Bevacizumab Plus Ixabepilone to Treat Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ravi A. Madan, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090057; 09-C-0057; NCT00820209 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Bevacizumab; Ixabepilone; Phase II
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bevacizumab with Ixabepilone (Experimental): Bevacizumab 15mg/kg every 3 weeks Ixabepilone given on days 1,2,3,4 and 5 of each three week cycle at a dose of 6mg/m(2)/day
  Interventions: Drug: Bevacizumab; Drug: Ixabepilone

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered intravenously every 3 weeks on an outpatient basis with the exception of admissions for the purpose of facilitating research studies. The dose of bevacizumab to be given is 15 mg/kg.
  Other Names: Avastin
Drug: Ixabepilone — Ixabepilone will be given on days 1, 2, 3, 4, and 5 of each three week cycle as a one hour intravenous infusion. The dose will be 6 mg/m(2)/day on five successive days.
  Other Names: Ixempra

SUMMARY:
Background:

* Substantial preclinical antitumor synergy supports the exploration of the combination of antiangiogenic compounds (including sunitinib and bevacizumab) plus ixabepilone. In Vivo, synergistic activity between ixabepilone and bevacizumab has been demonstrated using the 151-B human renal carcinoma xenograft model and this synergy compares favorably with other antiangiogenic inhibitors (i.e. sunitinib).
* Combination therapies of bevacizumab with chemotherapy demonstrated improved benefit compared with single-agent cytotoxics in multiple animal models and in humans.
* Clinical activity of both compounds used as single agents has been demonstrated in a broad spectrum of solid tumors. Bevacizumab and ixabepilone, when used as a single agent, have demonstrated substantial activity in renal cell carcinoma.
* Phase II studies with bevacizumab and ixabepilone suggest the absence of overlapping toxicities.
* Development of a well-tolerated and active bevacizumab/ixabepilone combination has the potential to further improve the treatment of metastatic renal cell carcinoma (mRCC), and could represent a second-line option after sunitinib or sorafenib are no longer of benefit or are intolerable.

Primary Objectives:

* Determine the objective response rate of the combination of ixabepilone and bevacizumab in patients with relapsed or refractory mRCC.
* Determine progression-free survival.
* Characterize the toxicity of the combination of ixabepilone and bevacizumab in patients with mRCC.
* Determine changes in biomarkers and evaluate correlation with clinical outcomes.

Eligibility:

* Pathologic confirmation of renal cell carcinoma (clear cell histology) by the Laboratory of Pathology, National Cancer Institute (NCI), or the Medical University of South Carolina.
* Presence of metastatic renal carcinoma, after progression or intolerance to Vascular endothelial growth factor receptor (VEGFR) inhibitors (sunitinib and/or sorafenib).
* Adequate organ and bone marrow function.

Design:

* Multi-center, open labeled phase II study
* Following a Simon two-stage optimal design, a maximum of 58 patients with metastatic RCC will be accrued.
* Ixabepilone will be administered daily as a one hour infusion on five successive days (daily x 5), every three weeks (one cycle equals 3 weeks or 21 days +/- 5 days). Following cycle 6, cycles will be spread out to 4 weeks or 28 days +/- 5 days. The starting dose will be a daily dose of 6 mg/m(2)/day, for a total per cycle dose of 30 mg/m(2).
* In addition, 15 mg/kg bevacizumab will be administered intravenously on day 1 of each cycle. The first infusion of bevacizumab will be 90 minutes in duration, the second 60 minutes in duration, and in all subsequent cycles bevacizumab will be infused over 30 minutes if prior infusions are well tolerated.

DETAILED DESCRIPTION:
Background:

* Substantial preclinical antitumor synergy supports the exploration of the combination of antiangiogenic compounds (including sunitinib and bevacizumab) plus ixabepilone. In Vivo, synergistic activity between ixabepilone and bevacizumab has been demonstrated using the 151-B human renal carcinoma xenograft model and this synergy compares favorably with other antiangiogenic inhibitors (i.e. sunitinib).
* Combination therapies of bevacizumab with chemotherapy demonstrated improved benefit compared with single-agent cytotoxics in multiple animal models and in humans.
* Clinical activity of both compounds used as single agents has been demonstrated in a broad spectrum of solid tumors. Bevacizumab and ixabepilone, when used as a single agent, have demonstrated substantial activity in renal cell carcinoma.
* Phase II studies with bevacizumab and ixabepilone suggest the absence of overlapping toxicities.
* Development of a well-tolerated and active bevacizumab/ixabepilone combination has the potential to further improve the treatment of metastatic renal cell carcinoma (mRCC), and could represent a second-line option after sunitinib or sorafenib are no longer of benefit or are intolerable.

Primary Objectives:

* Determine the objective response rate of the combination of ixabepilone and bevacizumab in patients with relapsed or refractory mRCC.
* Determine progression-free survival.
* Characterize the toxicity of the combination of ixabepilone and bevacizumab in patients with mRCC.
* Determine changes in biomarkers and evaluate correlation with clinical outcomes.

Eligibility:

* Pathologic confirmation of renal cell carcinoma (clear cell histology) by the Laboratory of Pathology, National Cancer Institute (NCI), or the Medical University of South Carolina.
* Presence of metastatic renal carcinoma, after progression or intolerance to vascular endothelial growth factor receptor (VEGFR) inhibitors (sunitinib and/or sorafenib).
* Adequate organ and bone marrow function.

Design:

* Multi-center, open labeled phase II study
* Following a Simon two-stage optimal design, a maximum of 58 patients with metastatic RCC will be accrued.
* Ixabepilone will be administered daily as a one hour infusion on five successive days (daily x 5), every three weeks (one cycle equals 3 weeks or 21 days +/- 5 days). Following cycle 6, cycles will be spread out to 4 weeks or 28 days +/- 5 days. The starting dose will be a daily dose of 6 mg/m(2)/day, for a total per cycle dose of 30 mg/m(2).
* In addition, 15 mg/kg bevacizumab will be administered intravenously on day 1 of each cycle. The first infusion of bevacizumab will be 90 minutes in duration, the second 60 minutes in duration, and in all subsequent cycles bevacizumab will be infused over 30 minutes if prior infusions are well tolerated.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects meeting all of the following criteria will be considered for enrollment into the study:

1. Pathologic confirmation of metastatic or unsectable renal cell carcinoma with predominant clear cell histology (greater than 70%) by the Laboratory of Pathology, National Cancer Institute (NCI) or the Medical University of South Carolina..
2. Progression on or after stopping treatment with an agent approved by the Food and Drug Administration (FDA) for the treatment of renal cell carcinoma (RCC). Patients must have received at least one FDA approved agent (axitinib, sunitinib, sorafenib, pazopanib, temsirolimus, interleukin-2 (IL-2), interferon or everolimus). Patients must be off prior IL-2 or interferon for 4 weeks prior to entry. They must be off sunitinib, sorafenib, pazopanib, axitinib, temsirolimus or everolimus or other tyrosine kinase inhibitor (TKIs) for 2 weeks prior to entry.
3. Eighteen years of age or older.
4. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
5. Resolution of any toxic effects of prior therapy (except alopecia) to NCI Common Terminology Criteria in Solid Tumors (CTCAE) v.3.0 through 12/31/10 and version 4.0 beginning 1/1/11 grade less than or equal to 1 and to baseline laboratory values as defined in inclusion criterion # 6.
6. Adequate organ and bone marrow function as evidenced by:

   * hemoglobin greater than or equal to 9.0 g/dL
   * absolute neutrophil count greater than or equal to 1.5 x 10(9)/L
   * platelet count greater than or equal to 100 x 10(9)/L
   * creatinine less than or equal to 1.5 times the ULN, OR measured creatinine clearance greater than or equal to 40 ml/min
   * urine proteinuria less than 20mg/dL on random protein creatinine ratio urine samples or a 24-hour urine protein less than 500 mg. NOTE: If on a random protein creatinine ratio the urine protein is greater that or equal to 20mg/dL, then obtain a 24 hour urine collection to accurately demonstrate that the 24 hour total is less than 500 mg/24 hours.
   * aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 times the upper limit of normal (ULN) (or less than or equal to 5 times the ULN if liver function abnormalities due to underlying malignancy)
   * total bilirubin less than or equal to 1.5 times the ULN
7. Subjects must be postmenopausal, surgically sterile, or using effective contraception. All female subjects of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days prior to enrollment. Effective contraception includes hormonal or barrier methods.
8. No other invasive malignancies within the past two years (with the exception of nonmelanoma skin cancers, non-invasive bladder cancer, stage I endometrial cancer or cervical cancer).
9. Subjects must agree to sign and date an Institutional Review Board (IRB)-approved subject informed consent form.
10. Subjects must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
11. Patients must have measurable disease either by conventional imaging or clinical examination.

EXCLUSION CRITERIA:

Subjects presenting with any of the following will not be included in the study:

1. Invasive procedures defined as follows:

   * Major surgical procedure, open biopsy or significant traumatic injury within 6 weeks prior to Day 1 therapy
   * Anticipation of need for major surgical procedures during the course of the study
   * Minor surgery, such as port-a-cath placement, and dental procedures, within 2 weeks.
   * (There will be no delay for percutaneous core biopsies or peripherally inserted central catheter (PICC)/internal jugular (IJ) line placement)
2. Cumulative radiation therapy to greater than 25% of the total bone marrow.
3. History of uncontrolled or labile hypertension, defined as blood pressure greater than 160/90 mm Hg (NCI CTCAE v.3.0 through 12/31/10 and version 4.0 beginning 1/1/11 grade greater than or equal to 2), on at least 2 repeated determinations on separate days within 15 days prior to study enrollment.
4. Any of the following within 6 months prior to study enrollment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class III or IV congestive heart failure; cerebrovascular accident or transient ischemic attack, grade greater than or equal to 2 peripheral neuropathy, peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, or other thromboembolic event.
5. Symptomatic spinal cord compression.
6. Evidence of clinically significant bleeding diathesis or underlying coagulopathy.
7. Antiretroviral therapy for human immunodeficiency virus (HIV) disease.
8. Pregnant (positive pregnancy test) or nursing women. Both fertile men and women must agree to use adequate contraceptive measures during study therapy and for at least 6 months after the completion of bevacizumab therapy.
9. Other severe acute or chronic medical or psychiatric condition, or significant laboratory abnormality requiring further investigation that may cause undue risk for the subjects safety, 18 inhibit protocol participation, or interfere with interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
10. Prior therapy with bevacizumab
11. Prior therapy with ixabepilone.
12. Patients on anticoagulant therapy will be evaluated on a case by case basis for inclusion.
13. Serious or non-healing wound, ulcer or bone fracture
14. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to day 1
15. Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
16. Known central nervous system (CNS) disease except for treated brain metastasis.

    -Treated brain metastases are defined as having no ongoing requirement for steroids and no evidence of progression or hemorrhage after treatment for at least 3 months, as ascertained by clinical examination and brain imaging (magnetic resonance imaging (MRI) or computed tomography (CT)). (Stable dose of anticonvulsants are allowed). Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, linear particle accelerator (LINAC), or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
17. Patients with known hypersensitivity of Chinese hamster ovary cell products or other recombinant human antibodies
18. Patients receiving cytochrome P450 3A4 (CYP3A4) inhibitors in section 3.6 that cannot be discontinued.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01-07 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ryan AM, Eppler DB, Hagler KE, Bruner RH, Thomford PJ, Hall RL, Shopp GM, O'Neill CA. Preclinical safety evaluation of rhuMAbVEGF, an antiangiogenic humanized monoclonal antibody. Toxicol Pathol. 1999 Jan-Feb;27(1):78-86. doi: 10.1177/019262339902700115. PMID 10367678
- [Background] Ferrara N, Chen H, Davis-Smyth T, Gerber HP, Nguyen TN, Peers D, Chisholm V, Hillan KJ, Schwall RH. Vascular endothelial growth factor is essential for corpus luteum angiogenesis. Nat Med. 1998 Mar;4(3):336-40. doi: 10.1038/nm0398-336. PMID 9500609
- [Background] Hellman S, Rosenthal DS, Moloney WC, Chaffey JT. The treatment of non-Hodgkin's lymphoma. Cancer. 1975 Aug;36(2):804-8. doi: 10.1002/1097-0142(197508)36:2+3.0.co;2-w. PMID 1157038
- [Result] Phase II clinicaltrial of bevacizumab plus ixabepilone in renal cell carcinoma. Mauricio Emmanuel Burotto Pichun, Nicolas Acquavella, Maureen Edgerly, Susan Elaine Bates, Sanjeeve Balasubramaniam and Antonio Tito Fojo; Journal of Clinical Oncology, 2014 Genitourinary Cancers Symposium (January 30 - February 1, 2014). Vol. 32, No 4_suppl (February 1 Supplement), 2014: 427
- [Derived] Burotto M, Edgerly M, Velarde M, Balasubramaniam S, Drabkin H, Gormaz JG, O'Sullivan C, Madan R, Fojo T. A Phase II Multi-Center Study of Bevacizumab in Combination with Ixabepilone in Subjects with Advanced Renal Cell Carcinoma. Oncologist. 2017 Aug;22(8):888-e84. doi: 10.1634/theoncologist.2017-0211. Epub 2017 Jul 5. PMID 28679644
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0057.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab With Ixabepilone
Started | 30
Completed | 5
Not Completed | 25
Not completed — Stopped treatment due to progression | 17
Not completed — Death | 1
Not completed — Discontinued treatment due to toxicities | 3
Not completed — Switched to alternative treatment | 2
Not completed — Refused further treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.17 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Prior Therapies [Median (Full Range); unit: therapies] | 2 [1 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: The time between the first day of treatment to the day of disease progression. Progression is defined by the Response Evaluation Criteria in Solid Tumors (RECIST). Progression is at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: up to 44 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 30
months | 8.3 [4.9 to 10.6]

2. Secondary Outcome: Number of Participants With an Objective Response (Complete Response (CR) or Partial Response (PR)) Per the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Response (complete response (CR) and partial response (PR)) was measured by the RECIST. Complete response is the disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: Two Years
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 30
Participants
  Complete Response | 0
  Partial Response | 3

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events, see the adverse event module. Adverse events are assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: Date treatment consent signed to date off study, approximately 84 months and 25 days
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 30
Participants | 30

4. Secondary Outcome: Number of Participants Who Had Biopsies
Description: To obtain tumor tissue and perform analysis for molecular changes in the tumor before and after a cycle of chemotherapy.
Time Frame: Baseline and Cycle 2 Day 1
Population: This outcome measure was not done because biopsy samples were not obtained.
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Time between the first day of treatment and the day of death.
Time Frame: Time between the first day of treatment and the day of death, assessed up to approximately 7 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 30
months | 15.0 [11.3 to 29.8]

6. Other Pre Specified Outcome: Protein Profiling of Vascular Endothelial Growth Factor A (VEGF-A), Vascular Endothelial Growth Factor Receptor 2 (VEGFR-2), Vascular Endothelial Growth Factor Receptor 3 (VEGFR-3), Beta Fibroblast Growth Factor (βFGF) and Erythropoietin From Baseline
Description: This assessment was intended as an exploratory analysis.
Time Frame: Cycle 1 Day 5 (C1D5), Cycle 2 Day 1 (C2D1), Cycle 4 and Cycle 6
Population: This outcome measure was not done. Data was not collected because the clinical data did not support further analysis and interest.
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Circulating Endothelial Cells (CECs)
Description: This assessment was intended as an exploratory analysis.
Time Frame: Baseline, Day 5, and Cycle 2 Day 1
Population: as for outcome 6
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Micro Vessel Density
Description: This assessment was intended as an exploratory analysis
Time Frame: Prior to cycle 2
Population: as for outcome 6
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Tumor Endothelial Markers (TEMs)
Description: This assessment was intended as an exploratory analysis.
Time Frame: Cycle 1 Day 5, Cycle 2 Day 1, Cycle 4 Day 1, and Cycle 6 Day 1
Population: as for outcome 6
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Growth Rate Constant (g)
Description: This assessment was intended as an exploratory analysis.
Time Frame: up to 50 days
Population: as for outcome 6
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Percentage of Participants With an Increase or Decrease in Forward Contrast Transfer Rate (Ktrans) Using MRI Versus Conventional Imaging
Description: This assessment was intended as an exploratory analysis.
Time Frame: Cycle 1 before day 1 of treatment and day 5 following infusion
Population: as for outcome 6
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Percentage of Participants With an Increase or Decrease in Reverse Contrast Transfer Rate (Kep) Using MRI Versus Conventional Imaging
Description: This assessment was intended as an exploratory analysis.
Time Frame: Cycle 1 before day 1 of treatment and day 5 following infusion
Population: as for outcome 6
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 0

13. Other Pre Specified Outcome: Regression Rate Constant (d)
Description: This assessment was intended as an exploratory analysis.
Time Frame: up to 50 days
Population: as for outcome 6
Arm/Group | Bevacizumab With Ixabepilone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 8Date treatment consent signed to date off study, approximately 4 months and 25 days
Arm/Group | Bevacizumab With Ixabepilone
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 9/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab With Ixabepilone (N=30)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (2)
Presyncope (Infections and infestations) | 1 (1)
Urinary tract obstruction (Nervous system disorders) | 1 (1)
Diarrhea (Renal and urinary disorders) | 1 (1)
Proteinuria (Gastrointestinal disorders) | 1 (1)
Stroke (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab With Ixabepilone (N=30)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Activated partial thromboplastin time prolonged (Investigations) | 16 (37)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (13)
Alkaline phosphatase increased (Investigations) | 8 (20)
Allergic reaction (Immune system disorders) | 2 (2)
Allergic rhinitis (Skin and subcutaneous tissue disorders) | 8 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (13)
Anal hemorrhage (Gastrointestinal disorders) | 1 (3)
Anemia (Blood and lymphatic system disorders) | 20 (180)
Anorexia (Metabolism and nutrition disorders) | 13 (26)
Anxiety (Psychiatric disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (14)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 9 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Blood and lymphatic system disorders - Other, bleeding gums and DVT (Blood and lymphatic system disorders) | 1 (2)
Blood bilirubin increased (Investigations) | 2 (2)
Blurred vision (Eye disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Bruising (Injury, poisoning and procedural complications) | 1 (2)
CPK increased (Investigations) | 4 (5)
Catheter related infection (Infections and infestations) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (22)
Creatinine increased (Investigations) | 18 (140)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 16 (35)
Dizziness (Nervous system disorders) | 5 (5)
Dry eye (Eye disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 9 (15)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Esophageal infection (Infections and infestations) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Fatigue (General disorders) | 2 (68)
Fever (General disorders) | 5 (5)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Gastrointestinal disorders - Other, excessive saliva (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hot flashes (Vascular disorders) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 9 (26)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 14 (52)
Hypermagnesemia (Metabolism and nutrition disorders) | 4 (7)
Hypernatremia (Metabolism and nutrition disorders) | 4 (9)
Hypertension (Vascular disorders) | 16 (479)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 (191)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (18)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 11 (32)
Hyponatremia (Metabolism and nutrition disorders) | 15 (48)
Hypophosphatemia (Metabolism and nutrition disorders) | 13 (26)
Hypotension (Vascular disorders) | 3 (5)
Hypothyroidism (Endocrine disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Infections and infestations - Other, lung (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (5)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Investigations - Other, bicarbonate low (Investigations) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 4 (5)
Lymphocyte count decreased (Investigations) | 17 (206)
Lymphocyte count increased (Investigations) | 2 (6)
Malaise (General disorders) | 1 (1)
Movements involuntary (Nervous system disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 5 (12)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (8)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Nail infection (Infections and infestations) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 12 (17)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 15 (42)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, basal cell (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nervous system disorders - Other, cold intolerance (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 13 (26)
Olfactory nerve disorder (Nervous system disorders) | 2 (2)
Pain (General disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 18 (33)
Platelet count decreased (Investigations) | 8 (40)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Presyncope (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 5 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rhinitis infective (Infections and infestations) | 2 (3)
Serum amylase increased (Investigations) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 2 (16)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (8)
Sinusitis (Infections and infestations) | 2 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (4) — 1 laceration; 1 scabs ; 2 ingrown toe nails
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2)
Somnolence (Nervous system disorders) | 2 (3)
Surgical and medical procedures - Other, knee replacement (Surgical and medical procedures) | 1 (1)
Syncope (Nervous system disorders) | 3 (4)
Thromboembolic event (Vascular disorders) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Upper respiratory infection (Infections and infestations) | 6 (8)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (14)
Watering eyes (Eye disorders) | 1 (1)
Weight loss (Investigations) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
White blood cell decreased (Investigations) | 15 (90)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2015-08-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT00923130/Prot_000.pdf